CLINICAL TRIAL: NCT01112852
Title: A Randomized, Controlled Trial of Ligation Plus Vasoconstrictor vs.Ligation Plus Proton Pump Inhibitor in the Control of Acute Esophageal Variceal Bleeding
Brief Title: EVL (Endoscopic Variceal Ligation) Plus Vasoconstrictor vs.Ligation Plus PPI( Proton Pump Inhibitor) in the Control of Acute Esophageal Variceal Bleeding
Acronym: EVL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Chairperson, National Science Council
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EVL + PPI; PPI for EVB (Other Grant/Funding Number: Taiwan National Science Council)
Record Dates: First submitted 2010-04-23; First posted 2010-04-28 (Estimated); Last update posted 2010-04-28 (Estimated); Status verified 2010-04

CONDITIONS: Esophageal Varices; Bleeding
Keywords: control of bleed
MeSH Terms: conditions — Esophageal and Gastric Varices; Hemorrhage | interventions — Somatostatin; Terlipressin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EVL + vasoconstrictor (Active Comparator): Somatostatin 6mg in 500 cc 5% dextrose, 250μg slow bolus IV infusion followed by 250μg per hour (6mg/ 24 hours) or Terlipressin 2mg bolus was instituted on enrollment followed by 1mg per 6 hours for 5 days. The use of either somatostatin or glypressin was at the discretion of doctors in charge.
  Interventions: Drug: somatostatin or terlipressin
- EVL + PPI (Experimental): Pantoloc 40 mg intravenously per day was instituted on enrollment and continued for 5
  Interventions: Drug: pantoloc 40 mg

INTERVENTIONS:
Drug: pantoloc 40 mg — pantoloc iv. infusion per day
  Other Names: pantoloc, a proton pump inhibitor
  Arms: EVL + PPI
Drug: somatostatin or terlipressin — Somatostatin 6mg in 500 cc 5% dextrose, 250μg slow bolus IV infusion followed by 250μg per hour (6mg/ 24 hours) or Terlipressin 2mg bolus was instituted on enrollment followed by 1mg per 6 hours for 5 days. The use of either somatostatin or glypressin was at the discretion of doctors in charge.
  Other Names: somatostatin and terlipressin are vasoconstrictors.
  Arms: EVL + vasoconstrictor

SUMMARY:
Previous studies showed that combination of endoscopic therapy with vasoconstrictor is better than either vasoconstrictor or endoscopic therapy alone in achieving the successful hemostatsis of acute variceal bleeding. The rationale of using vasoconstrictor is to enhance the efficacy of hemostasis by endoscopic therapy. Nowadays, endoscopic variceal ligation (EVL) has replaced endoscopic injection sclerotherapy (EIS) as the endoscopic treatment of choice in the arresting of acute esophageal variceal hemorrhage. EVL alone can achieve hemotasis up to 97% even in cases of active variceal hemorrhage. However, early rebleeding due to ligation-induced ulcer may be encountered. It appears that prevention of esophageal ulcers and bleeding by a proton pump inhibitor may be more logical than using a vasoconstrictor after cessation of bleeding by EVL.

DETAILED DESCRIPTION:
Previous studies showed that combination of endoscopic therapy with vasoconstrictor is better than either vasoconstrictor or endoscopic therapy alone in achieving the successful hemostatsis of acute variceal bleeding. The rationale of using vasoconstrictor is to enhance the efficacy of hemostasis by endoscopic therapy. Nowadays, endoscopic variceal ligation (EVL) has replaced endoscopic injection sclerotherapy (EIS) as the endoscopic treatment of choice in the arresting of acute esophageal variceal hemorrhage. EVL alone can achieve hemotasis up to 97% even in cases of active variceal hemorrhage. However, early rebleeding due to ligation-induced ulcer may be encountered. It appears that prevention of esophageal ulcers and bleeding by a proton pump inhibitor may be more logical than using a vasoconstrictor after cessation of bleeding by EVL.

Thus, we designed a controlled trial to compare the initial hemostasis, early rebleeding rate in cirrhotic patients presenting with acute variceal bleeding receiving either emergency EVL plus somatostatin infusion or losec infusion for 5 days.

AIMS:

To investigate whether the combination of EVL and somatostatin is superior to the combination of EVL and losec in terms of efficacy in the arresting of acute esophageal variceal bleeding and very early rebleeding.

ELIGIBILITY:
Inclusion Criteria:

* The etiology of portal hypertension is cirrhosis.
* Age ranges between 18-80 y/o.
* Patients presenting with acute esophageal variceal bleeding proven by emergency endoscopy within 12 hours. (Acute esophageal variceal bleeding was defined as: (1) when blood was directly seen by endoscopy to issue from an esophageal varix (active bleeding), or (2) when patients presented with red color signs on their esophageal varices with blood in esophagus or stomach and no other potential site of bleeding identified (inactive bleeding).
* EVL is performed after confirmation of acute esophageal variceal bleeding. Enrollment time: Immediately after EVL is completed and variceal bleeding is arrested.

Exclusion Criteria:

* Association with severe systemic illness, such as sepsis, COPD, uremia
* Association with gastric variceal bleeding
* Failure in the control of bleeding by emergency EVL
* Moribund patients, died within 12 hours of enrollment
* Uncooperative
* Ever received EIS, EVL within one month prior to index bleeding
* Child-Pugh's scores > 13

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2006-12; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Success rate of initial hemostasis | 5 days
  Definition of initial hemostasis Initial hemostasis was defined as achieving a 24h bleeding-free period within the first 48h after treatment together with stable vital signs based on Baveno consensus criteria.
  Very early rebleeding was defined as: UGI bleeding occurred after initial hemostasis and within 5 days after enrollment. UGI bleeding was proven to be from esophageal varices.
very early rebleeding | 48-120 hours after treatment
  Very early rebleeding is defined as episodes of variceal bleeding 48-120 hours after treatment.

SECONDARY OUTCOMES:
The amount of blood transfusion within 42 days | 42 days
  The amount of blood transfusion during admission was recorded.
Mortality | within 42 days
  Mortality within 42 days was recorded and compared.
The size and number of ulcers on varices | 2 weeks after treatment
  If p't agrees, a second look endoscopy is performed to detect ulcers.

CONTACTS AND LOCATIONS:
Overall Officials: Gin-Ho Lo, Principal Investigator — E-DA Hospital

REFERENCES:
- [Derived] Lo GH, Perng DS, Chang CY, Tai CM, Wang HM, Lin HC. Controlled trial of ligation plus vasoconstrictor versus proton pump inhibitor in the control of acute esophageal variceal bleeding. J Gastroenterol Hepatol. 2013 Apr;28(4):684-9. doi: 10.1111/jgh.12107. PMID 23278466